CLINICAL TRIAL: NCT06920654
Title: Stabilization of the Shoulder Joint Using a Latarjet-like Procedure.
Status: Enrolling by invitation | Type: Observational
Sponsor: Vestre Viken Hospital Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 774617
Record Dates: First submitted 2025-03-26; First posted 2025-04-10 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Shoulder Instability
Keywords: shoulder instability; recurrence; Latarjet; arthroscopy; bone block
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This retrospective cohort study aims to evaluate the clinical outcomes of patients who underwent arthroscopic shoulder stabilization using a bone block technique for chronic recurrent shoulder dislocations. The study will assess complications, reoperations, and functional outcomes measured by the Western Ontario Shoulder Instability (WOSI) score. Patients operated on within the past 1-8 years will be included. Data will be collected through structured telephone interviews and medical record reviews.

DETAILED DESCRIPTION:
Background Chronic recurrent shoulder dislocation presents a significant challenge in orthopedic surgery, with potential long-term consequences for patients' functionality and quality of life. Arthroscopic stabilization using a bone block harvested from the iliac crest, without screw fixation, is a relatively new technique designed to reduce the risk of recurrence by improving the anatomical integrity of the shoulder joint.

Indications for shoulder stabilization surgery with a bone graft, also known as the bone block procedure, are based on classical criteria considering both anatomical and functional aspects of shoulder instability. These criteria include recurrent anterior shoulder dislocations that do not respond to conservative treatment such as physical therapy, significant glenoid bone loss, Hill-Sachs lesions, or failed previous stabilization surgery, such as a Bankart repair, where patients continue to experience instability or recurrent dislocations. Bone block stabilization may also be indicated in patients with particularly high demands for shoulder function and stability, such as those engaged in activities or occupations with a high risk of shoulder dislocation.

The bone block procedure addresses these issues by transferring a segment of bone from the iliac crest to the glenoid defect, thereby increasing the articular surface area. Simultaneously, the anterior joint capsule is tightened and reinforced, and the infraspinatus tendon is secured into the Hill-Sachs defect (remplissage) to enhance shoulder stability. This procedure is typically performed when more conservative methods have failed to provide adequate stability or when the anatomical conditions of the shoulder suggest that other techniques are unlikely to yield satisfactory results.

This study aims to evaluate the long-term outcomes of this surgical method.

Objective The primary objective of this study is to evaluate the clinical outcomes of patients undergoing arthroscopic shoulder stabilization with a bone block for chronic recurrent shoulder dislocations. The focus will be on complications, reoperations, and functional outcomes assessed using the Western Ontario Shoulder Instability Index (WOSI).

Methods and Study Design This study will be a retrospective cohort study including patients who have undergone arthroscopic shoulder stabilization using the bone block technique.

Recruitment and Informed Consent Eligible patients will be identified through searches in electronic medical records. Patients will first receive an information letter about the study, followed by a phone call 1-2 weeks later, providing an opportunity to ask questions. If the patient consents to participate, a digital consent form will be sent. Once the patient has signed the consent form digitally, a follow-up phone interview will be scheduled to complete a structured questionnaire assessing functional outcomes and quality of life.

Data Collection Data will be collected through structured telephone interviews focusing on postoperative complications, reoperations, and functional outcomes. Additionally, medical records will be reviewed to obtain relevant operative details and preoperative data. Data collection will be conducted by independent observers.

Statistical Analysis Descriptive statistics will summarize patient characteristics, complications, and functional scores.

Paired t-tests or Wilcoxon rank-sum tests will compare pre- and postoperative WOSI and EQ-5D-5L scores.

Chi-square or Fisher's exact test will be used to analyze categorical data such as complication or reoperation rates.

Correlation and regression analyses will examine predictors of functional outcomes.

Statistical significance will be set at p < 0.05.

Ethical Considerations The study will be conducted in compliance with the Declaration of Helsinki and will require approval from the Regional Ethics Committee (REK) and the local institutional review board (PVO). All participants will provide informed consent, and patient data will be anonymized to ensure confidentiality.

Study Timeline The study is expected to commence in Fall 2024 and will run for approximately two years, with data collection and analysis planned from 2024 to 2026. Results will be published in peer-reviewed journals and presented at relevant orthopedic conferences.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgery for chronic recurrent shoulder dislocations.
* Surgery performed between 1-10 years before study inclusion.
* Patients aged 18 years or older who provide informed consent.

Exclusion Criteria:

* Patients with other concurrent shoulder surgeries unrelated to bone block stabilization.
* Patients with major orthopedic conditions affecting the study outcome.
* Patients with insufficient follow-up data.
* Patients who do not provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients who underwent arthroscopic shoulder stabilization with a bone block technique at a single orthopedic center. Approximately 40-50 patients are expected to be included, with a retrospective follow-up period of 1-10 years postoperatively.
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence | From the index surgery to the time of the telephone interview, which may be up to 10 years.
  Recurrence of shoulder instability (measured through patient-reported dislocation episodes).

SECONDARY OUTCOMES:
Postoperative complications | From the index surgery to the time of the telephone interview, which may be up to 10 years.
  Postoperative complications (documented in medical records and patient interviews).
WOSI score | At the time of the telephone interview, which may be up to 10 years after the index surgery.
  Functional shoulder outcomes assessed by the WOSI score.
HRQoL | At the time of the telephone interview, which may be up to 10 years after the index surgery.
  Health-related quality of life evaluated using EQ-5D-5L.

CONTACTS AND LOCATIONS:
Overall Officials: Per Reidar Høiness, MD Phd, Principal Investigator — Vestre Viken HF
Locations (1):
- Drammen Hospital, Drammen, Norway